CLINICAL TRIAL: NCT05831670
Title: An Early Phase 2 Clinical Study of KSP-0243 in Patients With Mild to Moderate Active Ulcerative Colitis
Brief Title: An Early Phase 2 Clinical Study of KSP-0243
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0243CT02
Record Dates: First submitted 2023-03-02; First posted 2023-04-26 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KSP-0243 (Experimental): Under double-blinding, KSP 0243 tablets will be orally administered.
  Interventions: Drug: KSP-0243
- Placebo (Placebo Comparator): Under double-blinding, placebo tablets will be orally administered.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KSP-0243 — Oral administration
  Arms: KSP-0243
Drug: Placebo — Oral administration
  Arms: Placebo

SUMMARY:
A phase 2a, randomized, double-blind, placebo-controlled, multicenter, parallel-group study to administer KSP-0243 or a placebo once daily after breakfast for 8 weeks in 100 patients with mild to moderate active ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 74 years old (both inclusive)
* Patients who have been given the diagnosis of ulcerative colitis for at least 12 weeks
* Patients with an endoscopic view typically seen with ulcerative colitis spreading > 15 cm from the anal verge
* Patients with mild to moderate active ulcerative colitis who meet the certain conditions
* Patients who have an inadequate response to a fixed-dose oral 5-ASA formulation (mesalazine or salazosulfapyridine) continued from at least 2 weeks prior to the start of the screening period

Exclusion Criteria:

* Patients who underwent an enterectomy or are expected to require an enterectomy during the study period (except appendectomy)
* Patients who have or suspected to have bacterium- or parasite-induced infectious enteritis (e.g., infection with Clostridium difficile)
* Patients with any of the following concomitant illnesses with the severity considered inappropriate as a study patient by the principal investigator or the subinvestigator or medical history thereof:
* Hepatic or renal disorders or cardiovascular, endocrine, metabolic, pulmonary, gastrointestinal, neurological, urological, genitourinary, and immune diseases,

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Clinical response rate based on the modified Mayo score at Week 8 | Up to 8 weeks
  The percentage of patients who satisfied both of the following requirements:
  * Decreases in the modified Mayo score by ≥ 30% and ≥ 2 points from baseline
  * The rectal bleeding subscore based on the Mayo score decreases by ≥ 1 point from baseline or the subscore becomes ≤ 1 point

SECONDARY OUTCOMES:
Clinical remission rate based on the modified Mayo score at Week 8 | Up to 8 weeks
  Clinical remission rate based on the modified Mayo score: The percentage of patients who satisfied all of the following requirements:
  * The stool frequency subscore based on the Mayo score is 0 or 1 point with no aggravation from baseline
  * The rectal bleeding subscore based on the Mayo score is 0 points
  * The endoscopy subscore of the Mayo score is 0 or 1 point
Clinical response rate based on the full Mayo score at Week 8 | Up to 8 weeks
  Clinical response rate based on the full Mayo score: The percentage of patients who satisfied all of the following requirements.
  * Decreases in the full Mayo score by ≥ 30% and ≥ 3 points from baseline
  * The rectal bleeding subscore based on the Mayo score decreases by ≥ 1 point from baseline or the subscore becomes ≤ 1 point
Clinical remission rate based on the full Mayo score at Week 8 | Up to 8 weeks
  Clinical remission rate based on the full Mayo score: The percentage of patients who satisfied all of the following requirements.
  * Full Mayo score is ≤ 2 points
  * All the subscores are ≤ 1 point
Incidence of adverse events (AE) and adverse drug reactions (ADR) | Up to 8 weeks
  - Adverse events, Adverse drug reactions
Laboratory tests (Hematology): Hemoglobin (g/dL) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory tests (Hematology): Hematocrit (%) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory tests (Hematology): Erythrocyte (10^10/L) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Hematology): Leukocyte (10^6/L) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Hematology): Neutrophil (10^8/L) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Hematology): Eosinophil (10^8/L) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Hematology): Basophil (10^8/L) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Hematology): Monocyte (10^8/L) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Hematology): Lymphocyte (10^8/L) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Hematology): Platelet (10^10/L) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Blood chemistry): Na (mEq/L) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Blood chemistry): K (mEq/L) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Blood chemistry): Cl (mEq/L) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Blood chemistry): Ca (mEq/L) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Blood chemistry): P (mEq/L) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Blood chemistry): Creatinine (mg/dL) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Blood chemistry): Total Bilirubin (mg/dL) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Blood chemistry): Direct Bilirubin (mg/dL) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Blood chemistry): Indirect Bilirubin (mg/dL) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Blood chemistry): Total Protein (g/dL) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Blood chemistry): Albumin (g/dL) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Blood chemistry): AST (U/L) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Blood chemistry): ALT (U/L) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Blood chemistry): γGTP (U/L) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Blood chemistry): ALP (U/L) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Blood chemistry): Creatinine kinase (U/L) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Blood chemistry): Uric acid (mg/dL) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Blood chemistry): BUN (mg/dL) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Blood chemistry): LDH (U/L) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Blood chemistry): Total Cholesterol (mg/dL) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Blood chemistry): Triglyceride (mg/dL) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Blood chemistry): Amylase (U/L) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Blood chemistry): Glucose (mg/dL) | Up to 8 weeks
  * Summary statistics, scattered plots before and after the dose will be presented.
  * Shift tables before and after dose will be presented.
Laboratory test (Urinalysis): Protein | Up to 8 weeks
  * Number and percentage of subjects will be presented.
  * Shift tables before and after the dose will be presented.
Laboratory test (Urinalysis): Glucose | Up to 8 weeks
  * Number and percentage of subjects will be presented.
  * Shift tables before and after the dose will be presented.
Laboratory test (Urinalysis): Urobilinogen | Up to 8 weeks
  * Number and percentage of subjects will be presented.
  * Shift tables before and after the dose will be presented.
Laboratory test (Urinalysis): Occult blood | Up to 8 weeks
  * Number and percentage of subjects will be presented.
  * Shift tables before and after the dose will be presented.
Vital signs: Systolic blood pressure (mmHg) | Up to 8 weeks
  - Summary statistics, scattered plots before and after the dose will be presented.
Vital signs: Diastolic blood pressure (mmHg) | Up to 8 weeks
  - Summary statistics, scattered plots before and after the dose will be presented.
Vital signs: Pulse rate (bpm) | Up to 8 weeks
  - Summary statistics, scattered plots before and after the dose will be presented.
Vital signs: Body temperature (°C) | Up to 8 weeks
  - Summary statistics, scattered plots before and after the dose will be presented.
Measured values and fluctuations in body weight | Up to 8 weeks
  - Body weight
ECG parameter: RR interval (msec) | Up to 8 weeks
  - Summary statistics will be presented for measured values and changes from baseline.
ECG parameter: PR interval (msec) | Up to 8 weeks
  - Summary statistics will be presented for measured values and changes from baseline.
ECG parameter: QRS interval (msec) | Up to 8 weeks
  - Summary statistics will be presented for measured values and changes from baseline.
ECG parameter: QT interval (msec) | Up to 8 weeks
  - Summary statistics will be presented for measured values and changes from baseline.
ECG parameter: QTcF interval (msec) | Up to 8 weeks
  - Summary statistics will be presented for measured values and changes from baseline.
ECG parameter: Pulse rate (bpm) | Up to 8 weeks
  - Summary statistics will be presented for measured values and changes from baseline.
KSP-0243 concentration in plasma at each time point | Up to 8 weeks
  - KSP-0243 concentration in plasma
KSP-0243 concentration in colorectal mucosa at Week 8 | Up to 8 weeks
  - KSP-0243 concentration in colorectal mucosa

CONTACTS AND LOCATIONS:
Overall Officials: Yoshitaka Shimizu, Study Director — Kissei Pharmaceutical Co., Ltd.
Locations (1):
- Research Site, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: No